CLINICAL TRIAL: NCT06485999
Title: Periodontal Outcomes and Digital Volumetric Variation Following BOPT Restorations
Acronym: BOPT
Status: Completed | Type: Observational
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Rubén Agustín-Panadero, Assistant Professor of Stomatology, University of Valencia
Other Study IDs: UV-INV_ETICA-3325009
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Teeth treated with the Biologically Oriented Preparation Technique (BOPT): No interventions will be administered.
  Interventions: Procedure: Biologically Oriented Preparation Technique

INTERVENTIONS:
Procedure: Biologically Oriented Preparation Technique — It is a preparation technique without a finish line, also known as the biologically oriented preparation technique (BOPT). In this protocol, the crown's anatomic emergence profile at the cementoenamel junction (CEJ) is eliminated with diamond rotary instruments to create a new prosthetic junction, adapted to the gingival margin. The aim of this protocol is to create a new anatomic crown with a prosthetic emergence profile that simulates the shape of the natural tooth.
  Other Names: Vertical tooth preparation.

SUMMARY:
Technology is becoming increasingly essential in dentistry, and many procedures now require the use of an intraoral scanner. The goal of scanning the oral cavity is to create digital impressions, which are crucial for the fabrication of any dental prosthesis, as three-dimensional models of the dentition are needed.

Alongside technological advancements, new techniques for preparation in fixed dental prosthetics are being developed. An example is the BOPT technique, which involves vertical tooth preparation without a finishing line, associated with gingival sulcus curettage. The technique aims to improve the health and stability of gingival tissues over time.

Since it is a technique still not widely used, there is a need to intensify studies on the subject, justifying the conduct of this observational research aimed at assessing, through scanning and image overlay programs, the volumetric change of gingival tissues after the installation of ceramic prostheses with BOPT-type carving

DETAILED DESCRIPTION:
The aim of this study was to analyze the behavior of the periodontal tissues around teeth in the anterior region when restored with zirconia single crowns, using a biologically oriented preparation technique (BOPT). The study will investigate tooth-supported single crowns in the anterior region that were fabricated with a full zirconia core, in 18 patients, in the past 3 years. Follow-up analysis will measure periodontal responses by evaluating the following variables: plaque index (PI); probing depth (PD); gingival index (GI); and gingival thickness adjacent to the restoration using intraoral scanning.

The images of the scanning before and after BOPT restoration will be overlap by using a software tool named Geomagic. This program can quantify the changes of gingival thickness in different points defined by the investigator.

ELIGIBILITY:
Inclusion Criteria:

* patients who had been treated previously by BOPT technique.
* patients aged over 18 years.

Exclusion Criteria:

* Cases where the scanners cannot be overlapping.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who have received prosthetic treatment at the Clinics of Odontology at the University of Valencia in the last 3 years, using the biological oriented preparation technique.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2024-03-02 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Gingival Volumetric Variation | May 2024
  Variation of gingival tickness following BOPT technique

SECONDARY OUTCOMES:
Plaque Index | May 2024
  Index of bacterial plaque
Probing Depth | May 2024
  Depht of gingival sulcus
Gingival Index | May 2024
  Index for measure the gingival inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Ruben A Panadero, PhD, Principal Investigator — University of Valencia
Locations (1):
- Universidad de Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://doi.org/10.1016/j.prosdent.2015.05.010